CLINICAL TRIAL: NCT03538769
Title: Acute Kidney Injury: Integrating E-alerts and Clinical Decision Support System to Improve Outcomes
Brief Title: AKI Management Using Electronic Alerts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Shina Menon, Assistant Professor, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000811
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline group (No Intervention): This will be the pre and post alert phase where e-alerts will not be sent to providers
- Alert group (Other): This will be the phase when e-alerts will be sent to the provider
  Interventions: Other: electronic alert and clinical decision support system

INTERVENTIONS:
Other: electronic alert and clinical decision support system — Providers taking care of patients will receive an electronic alert and will be guided to use a clinical decision support system
  Arms: Alert group

SUMMARY:
Acute kidney injury (AKI) is a common clinical event with severe consequences. In the United States alone, greater than one million hospitalized patients per year are diagnosed with AKI. It has been independently associated with prolonged hospital stays, 25-80% risk of in-hospital death, and future progression to chronic kidney disease. While there has been an increase in awareness about the prevalence and significance of AKI, studies have uncovered systematic failure in the management of AKI, largely relating to the failure of clinicians to recognize and manage the condition appropriately. This is where we can use electronic health records (EHRs) and electronic alerts (e-alerts) to our advantage. In this study, the investigators plan to use e-alerts integrated into a clinical decision support (CDS) system to improve the care of and outcomes of patients with AKI. The aims are to study the prevalence of AKI and its progression among hospitalized patients using an 'AKI sniffer' (an EHR based automated system) and to prospectively study if introducing a complex intervention (an e-alert combined with a clinical decision support system) will reduce progression of AKI in children. The investigators have developed an AKI care bundle which provides simple guidelines for management of AKI along with specific discharge instructions to improve follow up care. The primary outcome is AKI progression. Secondary outcomes include morbidity, mortality, length of hospital stay, need for renal replacement therapy, and recovery of renal function by time of hospital discharge. The investigators will also look at documentation of AKI and if these participants get appropriate follow up.

ELIGIBILITY:
Inclusion Criteria:

All patients between 6 months-18 years admitted to the surgical and medical floors of Seattle Children's Hospital

Exclusion Criteria:

1. History of chronic kidney disease stage 4 or worse (i.e., patients on chronic renal replacement therapy or glomerular filtration rate < 30 mL/min/1.73 m2)
2. History of renal transplantation within the last 3 months
3. History of nephrectomy within last 3 months
4. Patients admitted to observation units

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
AKI documentation | 28 days
  Documentation of AKI in progress notes and discharge summary

SECONDARY OUTCOMES:
AKI progression | 7 days
  Progression of AKI from Stage 1 to Stage 2/3

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menon S, Tarrago R, Carlin K, Wu H, Yonekawa K. Impact of integrated clinical decision support systems in the management of pediatric acute kidney injury: a pilot study. Pediatr Res. 2021 Apr;89(5):1164-1170. doi: 10.1038/s41390-020-1046-8. Epub 2020 Jul 3. PMID 32620006